CLINICAL TRIAL: NCT05214963
Title: Exploratory Clinical Study to Assess Tolerability, Safety, and Response to Non-invasive Peripheral Nerve Stimulation (NPNS) in Medication-naïve and Medication-refractory Restless Legs Syndrome (RLS) Patients
Brief Title: Noninvasive Peripheral Nerve Stimulation for Medication-Naive and Medication-Refractory RLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noctrix Health, Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT-02; R44NS117294 (NIH)
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 between Active treatment and Sham control
Who Masked: Participant
Masking Description: Single-blind [Participant]
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active neurostimulation (Active Comparator): Noninvasive peripheral nerve stimulation device programmed to deliver active stimulation
  Interventions: Device: NTX100 Neuromodulation System - Active
- Sham neurostimulation (Sham Comparator): Noninvasive peripheral nerve stimulation device programmed to deliver non-therapeutic (sham) stimulation
  Interventions: Device: NTX100 Neuromodulation System - Sham

INTERVENTIONS:
Device: NTX100 Neuromodulation System - Active — Noninvasive peripheral nerve stimulation device programmed to active mode
  Arms: Active neurostimulation
Device: NTX100 Neuromodulation System - Sham — Noninvasive peripheral nerve stimulation device programmed to sham mode
  Arms: Sham neurostimulation

SUMMARY:
Prospective multi-site randomized sham-controlled study evaluating tolerability and efficacy of noninvasive peripheral nerve stimulation (NPNS) for patients with moderate-severe primary Restless Legs Syndrome (RLS) who are either medication-naive or medication-refractory.

DETAILED DESCRIPTION:
The study consists of a series of two 2-week phases:

Phase 1: Baseline evaluation of RLS and sleep Phase 2: Prospective, single-blinded, 1:1 randomized evaluation of response to NPNS treatment (Active treatment: Sham control)

Additionally, subjects will have the option to consent to a third phase, which includes overnight polysomnography (PSG) evaluation of sleep with Active treatment and with no treatment (baseline), in randomized order.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has received a medical diagnosis of primary restless legs syndrome (RLS).
2. Subject is either medication-naïve or medication-refractory.
3. Subject has moderate-severe RLS symptoms as defined by a score of 15 or greater points on IRLS (International Restless Legs Syndrome Study Group Rating Scale) over the week prior to study entry.
4. RLS symptoms interfered with sleep on at least 3 nights per week during the month prior to study entry.
5. RLS symptoms are most significant in the subject's lower legs and/or feet.
6. RLS symptoms are most significant after 6pm.
7. Subject agrees to not change dosage or schedule of any medications that are known to impact RLS symptoms during the study, including RLS medications, antidepressants, sleep medications, or sedative antihistamines.
8. Subject agrees to not make major lifestyle changes during the study that would significantly affect bedtime, such as major changes to diet, exercise, or career.
9. Subject possesses the necessary equipment, internet/phone accessibility, and communication ability to complete electronic questionnaires and respond to electronic communications and phone calls from the research staff throughout the in-home portion of the study.
10. Subject is ≥ 22 and ≤ 89 years of age when written informed consent is obtained.
11. Subject has signed a valid, IRB-approved informed consent form, can understand the requirements of the study and instructions for device usage, and can converse in English.

Exclusion Criteria:

1. Subject has RLS that is known to be caused by another diagnosed condition (i.e. secondary RLS).
2. Subject is taking an unstable or inconsistent dose or schedule of medication that is likely to impact RLS symptoms, such as antidepressants, sleep medications, or sedative antihistamines or has changed dosage within the past 30 days.
3. Subject has changed dose and schedule of RLS medications within the month prior to study entry or is otherwise on an inconsistent dose or schedule of RLS medications.
4. Subject has prior experience with Noctrix Health NPNS devices.
5. Subject was misdiagnosed with RLS, as determined by the investigator (e.g. actual diagnosis of PLMD, arthritis, leg spasms or neuropathy without comorbid RLS).
6. Subject has a primary sleep disorder other than RLS that significantly interferes with sleep at the present time (e.g. obstructive sleep apnea stably controlled via CPAP would not be an exclusion).
7. Subject has active medical device implant anywhere in the body (including but not limited to pacemakers, spinal cord stimulators, deep brain stimulators) or metal implant at the site of study device electrode application.
8. Subject has severe peripheral neuropathy affecting the lower legs and/or subject has neuropathy and is unable to clearly distinguish between symptoms of neuropathy and symptoms of RLS.
9. Subject has been diagnosed with one of the following conditions:

   * Epilepsy or other seizure disorder
   * Current, active or acute or chronic infection other than common cold
   * A malignancy within the past 5 years (not including basal or squamous cell skin cancer)
   * Stage 4-5 chronic kidney disease or renal failure
   * Severe movement disorder symptoms (Parkinson's disease, Huntington's disease, dyskinesia, dystonia)
   * Deep vein thrombosis
   * Multiple sclerosis
10. Subject has moderate or severe cognitive disorder or mental illness.
11. Subject has current diagnosis of iron-deficient anemia or history of iron-deficient anemia within the past year.
12. Subject has known allergy to device materials or severe previous reaction to medical adhesives or bandages.
13. Subject has severe edema affecting lower legs.
14. Subject has any of the following at or near the location of device application.

    * Acute injury
    * Cellulitis
    * Open sores
    * Other skin condition
15. Subject is on dialysis or anticipated to start dialysis while participating in the study
16. During the NTX100 calibration process, which is identical for subjects in the active and sham arms, subject reports not feeling stimulation sensations up to an intensity of 30mA, the subject finds stimulation intensities less than 15 mA to be uncomfortable or distracting, or the device does not properly fit the subject.
17. Subject has received an investigational drug or device within the last 30 days or is planning to receive an investigational device during the duration of the study.
18. Subject is pregnant or trying to become pregnant.
19. Subject has undergone a major surgery (excluding dental work) in the previous 30 days.
20. Subject is unable or unwilling to comply with study requirements.
21. Subject has another medical condition that may put the subject at risk as determined by the investigator.
22. Subject has another medical condition that may affect validity of the study as determined by the investigator.

Ages: 22 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Tolerability based on Withdrawal Rate | 2 weeks
  Percentage of subjects who withdraw from study citing lack of tolerability of the study device as the primary reason for withdrawal
Actigraphy-Based Sleep Efficiency | 1 week
  The ratio of wake after sleep onset to total sleep time, as measured by actigraphy
Actigraphy-Based Total Sleep Time | 1 week
  Total sleep duration, as measured by actigraphy

SECONDARY OUTCOMES:
Frequency of Device Usage | 2 weeks
  The frequency of study device usage on nights with RLS symptoms
Grade 2 or higher device-related adverse events | 2 weeks
  Frequency of Grade 2 or higher device-related adverse events
Grade 3 or higher device-related adverse events | 2 weeks
  Frequency of Grade 3 or higher device-related adverse events
Polysomnography-Based Sleep Efficiency | 1 night
  The ratio of wake after sleep onset to total sleep time, as measured by polysomnography
Polysomnography-Based Total Sleep Time | 1 night
  Total duration of sleep, as measured by polysomnography
International Restless Legs Syndrome Study Group Rating Scale (IRLS) score | 1 week
  IRLS is a participant-rated questionnaire that rates RLS severity from 0-40, where 40 is the most severe
Patient Global Impressions of Improvement Responder Rate | 1 week
  Percentage of subjects with a Patient Global Impressions of Improvement (PGI-I) rating of Much Improved or Very Much Improved
Polysomnography-Based Percentage of Stage 3 Sleep | 1 night
  Mean percentage of total sleep time in Stage 3 sleep, as measured by polysomnography
Polysomnography-Based Percentage of REM Sleep | 1 night
  Mean percentage of total sleep time in REM sleep, as measured by polysomnography

OTHER OUTCOMES:
Medical Outcomes Study Sleep Problems Index II (MOS-II) score | 2 weeks
  MOS-II is a subscale of the participant-rated MOS questionnaire that measures subjective sleep quality.
Medical Outcomes Study Sleep Problems Index I (MOS-I) score | 2 weeks
  MOS-I is a subscale of the participant-rated MOS questionnaire that measures subjective sleep quality.
Actigraphy-Based Sleep Onset Latency | 2 weeks
  Time to fall asleep, as measured by actigraphy
Polysomnography-Based Sleep Onset Latency | 1 night
  Time to fall asleep, as measured by polysomnography
Polysomnography-Based Percentage of Stage 2 Sleep | 1 night
  Mean percentage of total sleep time in Stage 2 sleep, as measured by polysomnography
Numerical Rating Scale in Suggested Immobilization Test at 30 minutes | 30 minutes
  Rating of severity of RLS symptoms in Suggested Immobilization Test
Numerical Rating Scale in Suggested Immobilization Test at 60 minutes | 60 minutes
  Rating of severity of RLS symptoms in Suggested Immobilization Test
Numerical Rating Scale in Suggested Immobilization Test at 90 minutes | 90 minutes
  Rating of severity of RLS symptoms in Suggested Immobilization Test

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Charlesworth, PhD, Study Director — Noctrix Health, Inc.
Locations (3):
- United States (3):
  - SRI International Human Sleep Research Lab, Menlo Park, California
  - Sleep Medicine Specialists of California, San Ramon, California
  - Clayton Sleep Institute, St Louis, Missouri